CLINICAL TRIAL: NCT07081308
Title: Clinical Evaluation of a Brain-computer Interface Integrated With Plantar Pneumoorthoses for Motor and Cognitive Rehabilitation in Stroke Survivors
Brief Title: Brain-computer Interface With Plantar Pneumoorthoses for Post-stroke Rehabilitation
Acronym: BRAIN-WALK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center of Neurology, Russia (Other Government)
Collaborators: Pirogov Russian National Research Medical University (Other); Institute of Higher Nervous Activity and Neurophysiology of RAS (Unknown)
Responsible Party: Principal Investigator, Natalia Suponeva, Director of Institute, Research Center of Neurology, Russia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIRS-BCI-Korvit
Record Dates: First submitted 2025-07-08; First posted 2025-07-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Brain-computer interface; Near infrared spectroscopy; gait recovery; stroke rehabilitation; Neurobiofeedback
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCI (Experimental): Stroke patients receiving NIRS-BCI-pneumoorthesis training in combination with standard therapy
  Interventions: Device: NIRS-BCI-pneumoorthesis
- Control (No Intervention): Stroke patients receiving standard therapy

INTERVENTIONS:
Device: NIRS-BCI-pneumoorthesis — Patients recieve 10 NIRS-BCI-pneumoorthesis trainings of 16 minutes each over 2 weeks.
  NIRS-BCI-pneumoorthesis Components: NIRScout hardware-software complex (16 light sources, 8 detectors); Software for brain activity classification; Korvit system for plantar support load reproduction; 22-inch monitor for task demonstration.
  Training Procedure: Patient seated with lower limbs fixed in pneumatic orthoses; Task: kinesthetically imagine walking or relax; Feedback: visual (color change on screen) and tactile (support load through orthosis).
  Training structure: 16 blocks alternating walking imagination and relaxation
  Other Names: neurobiofeedback
  Arms: BCI

SUMMARY:
STUDY PURPOSE The investigators are testing a new rehabilitation system that helps stroke patients recover their ability to walk and think more clearly. This system, called brain-computer interface with plantar pneumorthoses, uses brain signals to control a special device that provides gentle pressure to the feet, similar to what you feel when walking. The goal is to help patients regain walking skills, improve memory and thinking, and feel better emotionally.

STUDY QUESTIONS

The main questions the study aims to answer are:

Whether the investigated technology can improve walking in post-stroke patients? Whether the training to control the technology can improve cognitive function in post-stroke patients?

HOW THE STUDY WORKS The investigators compare two groups - one using the new system, another group receiving standard rehabilitation therapy.

Up to 15 patients will try the new system: 10 sessions, each lasting 12 minutes (about 2 weeks, Monday-Friday).

WHAT HAPPENS DURING TREATMENT?

The equipment includes:

Brain monitoring device: Safe infrared light sensors placed on the patient's head (like a cap) Computer software: Reads brain signals when the patient thinks about walking Foot device: Special pneumatic shoes that provide gentle pressure to the patient's feet Screen: Shows visual feedback during training.

What the patient will do:

Sit comfortably in a chair with special shoes on their feet, Complete the task: imagine walking or relax when instructed, What the patient will experience: They will see colors change on the screen and feel gentle pressure on their feet.

DETAILED DESCRIPTION:
INTERVENTION NIRS-BCI-Korvit System Components: NIRScout hardware-software complex (16 light sources, 8 detectors); Software for brain activity classification; Korvit pneumoorthesis for plantar support load reproduction; 22-inch monitor for task demonstration Training Procedure: Patient seated with lower limbs fixed in pneumatic orthoses; Task: kinesthetically imagine walking or relax; Feedback: visual (color change on screen) and tactile (support load through orthosis).

Training structure: 16 blocks alternating walking imagination and relaxation/ ASSESSMENT

Motor Function:

* Fugl-Meyer Scale for Lower Extremity (maximum 34 points, clinically significant improvement ≥6 points);
* 10-meter Walk Test (clinically significant improvement ≥0.16 m/s);
* Timed Up and Go Test (clinically significant improvement ≥3 seconds).

Cognitive Functions and Emotional State:

* Addenbrooke's Cognitive Examination III (ACE III);
* Hospital Anxiety and Depression Scale (HADS). EXPECTED OUTCOMES.

The study aims to confirm the effectiveness of NIRS-BCI combined with plantar support load simulator for:

* Gait restoration;
* Cognitive function improvement;
* Emotional state normalization in post-stroke patients SAFETY The procedure is safe and poses no health risks. Possible minor fatigue after sessions. The study can be discontinued at any stage upon patient request or if adverse effects occur.

INNOVATION This research represents a novel approach combining non-invasive brain-computer interface technology with proprioceptive feedback systems for comprehensive post-stroke rehabilitation, addressing both motor and cognitive recovery simultaneously

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Primary or recurrent supratentorial ischemic stroke
* Stroke onset 7 days to 24 months
* Moderate to mild post-stroke lower limb motor impairments
* Clinical stability
* Voluntary participation and signing of informed consent

Exclusion Criteria:

* Severe cognitive impairments preventing instruction compliance
* Sensory or severe motor aphasia
* Severe visual impairments
* Lower limb contractures
* Inability to maintain sitting position

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Walking speed change as assessed by the 10-Meter Walk Test | From enrollment to the end of treatment at 2 weeks
  Before and after treatment course
Lower extremity functional improvement as assessed by the Fugl-Meyer Assessment | From enrollment to the end of treatment at 2 weeks
  Before and after treatment course

SECONDARY OUTCOMES:
Lower extremity functional improvement as assessed by the Timed Up and GO test | From enrollment to the end of treatment at 2 weeks
  Before and after treatment course
Cognitive function improvement as assessed by the Addenbrooke's cognitive examination - III | "From enrollment to the end of treatment at 2 weeks
  Before and after treatment course

OTHER OUTCOMES:
Emotional improvement as assessed by the Hospital Anxiety and Depression Scale | From enrollment to the end of treatment at 2 weeks
  Before and after treatment course

CONTACTS AND LOCATIONS:
Locations (1):
- Russian center of Neurology and Neurosciences, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No